CLINICAL TRIAL: NCT03626675
Title: Anterior Segment Changes Before and After Uneventful Combined Phaco-Trabeculectomy by Using Optical Coherence Tomography (OCT)
Brief Title: Anterior Segment Changes by Optical Coherence Tomography (OCT) in Phaco- Trabeculectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, shymaa kamel Ibrahim Hady, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ASCBAPTBUOCT
Record Dates: First submitted 2018-08-07; First posted 2018-08-13 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-08

CONDITIONS: Angle Closure Glaucoma; Glaucoma; Cataract Secondary
MeSH Terms: conditions — Glaucoma, Angle-Closure; Glaucoma; Capsule Opacification

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Other): They will be subjected to:
  Preoperative A-complete ophthalmic examination will be done for every patient; B- Biometric parameters measured with the AS-OCT C- Medical fitness for all patients D- Informed consent will be obtained from all patients after through explanation of operation and its potential benefits and risks.
  Surgery combined Phaco trabeculectomy
  Post operative:
  -Follow-up examinations will be performed for every patient at 1day, 1 week, 1 and 3 months postoperatively.
  and biometric parameters measured with the AS-OCT before and after the surgery will be used to collect the data.
  -The data will be managed and analysed with confidentiality by scientifically qualified persons
  Interventions: Procedure: phaco- trabeculectomy

INTERVENTIONS:
Procedure: phaco- trabeculectomy — combined phaco-trabeculectomy surgery

SUMMARY:
1. Develop a measurement protocol by OCT imaging and characterization of the anterior chamber change in glaucoma patients before and after surgery.
2. Show the effect of combined surgery in control of intra ocular pressure.

DETAILED DESCRIPTION:
Definitions Glaucoma represents a group of diseases defined by a characteristic optic neuropathy that is consistent with excavation and undermining of the neural and connective tissue elements of the optic disc and by the eventual development of distinctive patterns of visual dysfunction .Pre-perimetric glaucoma is a term that is sometimes used to denote glaucomatous changes in the optic disc in patients with normal visual fields.

Glaucoma and cataract incidence increases with age. Special considerations are needed when choosing which surgical strategy to undertake when either of these two conditions requires surgical management. When performed prior to cataract surgery, trabeculectomy increases the risk of cataract formation by up to 78%, while subsequent cataract surgery may increase the risk of elevated intraocular pressure or trabeculectomy failure. By contrast, when cataract surgery alone is performed in glaucoma patients; an early postoperative intraocular pressure spike sometimes requiring medical treatment is commonly reported. Therefore, phacotrabeculectomy, a procedure that combines the management of these two conditions together in one surgery, may be considered in these situations.

When to Consider Combined Surgery

Combined cataract extraction and glaucoma surgery (trabeculectomy, glaucoma drainage implant surgery, or any of the newer surgical approaches for glaucoma) should be carefully selected and individualized depending on clinical findings in each case:

* Cataract surgery alone is sufficient for patients with well controlled in intraocular pressure in the setting of early to moderate optic nerve damage.
* Patients with uncontrolled intraocular pressure in the presence of severe optic nerve damage should receive glaucoma surgery first, followed by cataract extraction a few months later
* Combined surgery may be best suited for a patient with a visually significant cataract with uncontrolled glaucoma despite maximal medical therapy and/or laser trabeculoplasty. Cost is often an issue for many patients and eliminating medications can help reduce the financial burden. Poor compliance with glaucoma medications can also be an issue to consider both procedures together.

The indication for phaco-trabeculectomy was the simultaneous presence of a visually significant cataract and open angle glaucoma requiring medications, poor patient compliance, advanced glaucomatous optic nerve damage or visual field loss, or medically uncontrolled glaucoma.

Effect of cataract surgery on anterior segment:

Cataract surgery and intraocular lens implantation lead to significant increases in anterior chamber depth and anterior chamber angle.

Trabeculectomy lead to significant decrease in anterior chamber depth and anterior chamber angle.The effects of trabeculectomy on anterior segment parameters measured by optical biometry in Primary open-angle glaucoma and pseudoexfoliation glaucoma and found in primary open angle glaucoma , intraocular pressure and anterior chamber depth decreased at the 1st and 3rd months significantly. Conclusion: Trabeculectomy cause some differences in anterior segment parameters in both primary open angle glaucoma and pseudoexfoliation cases and the differences between these changes in both groups were found to be insignificant.

Anterior Segment - Optical Coherence Tomography is a useful tool to evaluate filtering blebs or glaucoma drainage devices in the postoperative period. Clinically , blebs can be described as diffuse, cystic, encapsulated, or flat. However, these descriptions are subjective and there may be cases in which clinical appearance does not correlate with bleb function. Therefore, visualizing intra bleb morphology with anterior segment imaging may enhance our understanding of different surgical outcomes and wound healing. The noncontact anterior Segment - Optical Coherence Tomography scanning provides a significant advantage over ultrasound biomicroscopy in eliminating direct trauma to the bleb or reducing the risk of potential infection that could occur with the use of an eye-cup or probe .In addition, the higher scanning resolution of allows differentiating the subconjunctival fluid collection and the supra sclera fluid space. The anterior segment - optical coherence tomography used to describe intra- bleb morphology and structures, including bleb wall thickness, subconjunctival fluid collections, supra sclera fluid space, sclera flap thickness, and intra-bleb intensity. Anterior segment - optical coherence tomography allows visualization of the glaucoma drainage devices in the anterior chamber to assess their position or potential occlusion .

Effect of phacotrabeculectomy on anterior chamber depth:

Phacotrabeculectomy lead to increases in anterior chamber depth and anterior chamber angle. Poon, Linda Yi-Chieh et al studied comparison of surgical outcomes after phacotrabeculectomy in primary angle-closure glaucoma versus primary open-angle glaucoma found; the primary angle closure glaucoma group had an anterior chamber depth that was significantly shallower than the primary open-angle glaucoma group prior to surgery. However, after surgery, the mean anterior chamber depth in the primary angle closure glaucoma group increased to a depth similar to the primary open-angle glaucoma group.

Imaging of the anterior segment of the eye Imaging of the anterior segment of the eye offers an objective method for visualizing the angle and adjacent anatomical structures. In addition to qualitative analyses, some imaging modalities permit quantitative analyses that can be used to monitor change or progression over time.

Ultrasound Biomicroscopy uses high frequency ultrasound (35-100 MHz) to provide high resolution images of the angle. Ultrasound Biomicroscopy has shown good agreement with gonioscopy in assessing the anterior chamber angle. Although is a useful technology capable of providing both qualitative and quantitative analyses, its major advantage lies in its ability to visualize structures posterior to the iris to detect various causes of secondary angle closure, such as plateau iris, ciliary effusions, or irido-ciliary masses. The disadvantages of ultrasound biomicroscopy include required supine position, use of anesthesia, need for a skilled examiner, longer image acquisition time, and contact with the eye using a cup with a coupling medium or a probe that can lead to corneal abrasion or potential infection.

Anterior Segment Optical Coherence Tomography uses the principle of low-coherence interferometry instead of ultrasound to produce, cross sectional, non-contact, three-dimensional, high-resolution imaging modality of the anterior segment of the eye. The technique measures the delay and intensity of the light reflected from the tissue structure being analyzed and compares it with the light reflected by a reference mirror. The combination of these two signals results in interference phenomenon. The signal intensity depends on the optical properties of the tissues, and the device uses these signals to construct a sagittal cross-section image of the structure being analyzed. OCT technology was initially used to produce images of the posterior segment of the eye by using a wavelength of 820nm. In 2001, the wavelength was altered to 1310nm to allow better penetration through light retaining tissues such as the sclera and limbus and to improve visualization of the anterior segment. Compared with ultrasound biomicroscopy , this technology provides a higher axial resolution and faster sampling rate (2.0 kHz versus 0.8 kHz). Another main clinical advantage over ultrasound biomicroscopy is its ability to provide non contact scanning in a seated, upright position..The major drawback for anterior segment optical coherence tomography is its inability to visualize structures posterior to the iris due to blockage of wavelength by pigment. This limits its application in screening several secondary causes of angle closure, such as plateau iris, ciliary body cyst or tumor, lens subluxation, or ciliary effusions.

Biometric parameters which can be measured with the anterior segment optical coherence tomography:

Iris thickness ,iris cross- sectional area ,iris curvature ,AC depth ,AC width ,angle opening distance , angle recess area , scleral thickness, trabecular meshwork ciliary process distance ,trabecular iris angle , lens vault.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* Diagnosed primary open angle glaucoma
* Visual field defects and optic nerve head appearance characteristic for glaucoma
* Angle closure predisposition as evidenced from gonioscopy.
* Neovascularization in the anterior chamber angle
* pseudo-exfoliation glaucoma as evidenced from slit lamp examination
* No cataract surgery.
* No glaucoma surgery
* No degenerative changes in the retina in funduscopy after mydriasis

Exclusion Criteria:

* -previous glaucoma surgery
* Previous cataract surgery
* Presence of any abnormalities preventing reliable measurements
* Ocular inflammation and ocular disease interfering with the study
* Corneal, macula, and other corneal disease.
* No fixation Funds lesions such as diabetic retinopathy or retinal detachment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-15 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Biometric parameters measured with the AS-OCT (AC depth (ACD)) after surgery. - anterior chamber depth in mm | one week post operative
  anterior chamber depth in mm Distance from corneal endothelium to anterior surface of the lens

SECONDARY OUTCOMES:
other biometric parameters measured with the AS-OCT, | 1,3,6, month postoperative
  Parameter Unit
  Iris thickness μT Iris curvature μC AC width μC Angle opening distance μO Angle recess area μR Trabecular iris angle Degrees Lens vault μV
intra ocular pressure | 1,3,6, month postoperative
  intra ocular pressure in mm hg

CONTACTS AND LOCATIONS:
Overall Officials: Omar M Ali, MD,professor, Study Director — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Salim S. The role of anterior segment optical coherence tomography in glaucoma. J Ophthalmol. 2012;2012:476801. doi: 10.1155/2012/476801. Epub 2012 Aug 1. PMID 22900146
- [Result] Maslin JS, Barkana Y, Dorairaj SK. Anterior segment imaging in glaucoma: An updated review. Indian J Ophthalmol. 2015 Aug;63(8):630-40. doi: 10.4103/0301-4738.169787. PMID 26576519
- [Result] Sharma R, Sharma A, Arora T, Sharma S, Sobti A, Jha B, Chaturvedi N, Dada T. Application of anterior segment optical coherence tomography in glaucoma. Surv Ophthalmol. 2014 May-Jun;59(3):311-27. doi: 10.1016/j.survophthal.2013.06.005. Epub 2013 Oct 15. PMID 24138894
- [Result] Hong CJ, Trope GE. Glaucoma. CMAJ. 2015 Sep 8;187(12):E398-9. doi: 10.1503/cmaj.140401. Epub 2014 Nov 24. No abstract available. PMID 25421984